CLINICAL TRIAL: NCT03126188
Title: Study of the Effect of Antidepressant Drugs on Neurotrophic Factors in Patients With Depression
Status: Completed | Type: Observational
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, BISWA RANJAN MISHRA, Associate Professor, All India Institute of Medical Sciences, Bhubaneswar
Other Study IDs: T/IM-F/Psych/15/20
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Depressive Episode
MeSH Terms: interventions — Sertraline; Dothiepin; Venlafaxine Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Sertraline group: Mild and Moderate depressive episode without somatic syndrome who are treated with Sertraline. Tab. Sertraline 50 mg/day, which will be optimized to 75mg/day after 2 weeks if required, and maintained on the same dose for a minimum period of 6 weeks.
  Interventions: Drug: Sertraline
- Dosulepin group: Mild and Moderate depressive episode with somatic syndrome who were treated with Dosulepin. Tab. Dosulepin 25mg/day, which will be gradually hiked up to 75mg/day over 2 weeks
  Interventions: Drug: Dosulepin
- Venlafaxine group: Severe depressive episode without psychotic symptoms who were treated with Venlafaxine. Tab. Venlafaxine 75mg/day, which will be hiked to 112.5 mg/day after 2 weeks, and the patients will be continued on the same dose for a minimum period of 6 weeks.
  Interventions: Drug: Venlafaxine

INTERVENTIONS:
Drug: Sertraline — Tab. Sertraline 50 mg/day, which will be optimized to 75mg/day after 2 weeks if required, and maintained on the same dose for a minimum period of 6 weeks.
  Groups: Sertraline group
Drug: Dosulepin — Tab. Dosulepin 25mg/day, which will be gradually hiked up to 75mg/day over 2 weeks,and the patients will be continued on the same dose for a minimum period of 6 weeks.
  Groups: Dosulepin group
Drug: Venlafaxine — Tab. Venlafaxine 75mg/day, which will be hiked to 112.5 mg/day after 2 weeks, and the patients will be continued on the same dose for a minimum period of 6 weeks.
  Groups: Venlafaxine group

SUMMARY:
The aim of the present study will be to observe the changes in the NTs like Nerve growth factor, Neurotrophin-3, and Neurotrophin-4 in patients with depression and study the effect of various antidepressants like Sertraline (SSRI), Dosulepin (TCA), and Venlafaxine (SNRI) on their levels.

DETAILED DESCRIPTION:
Depression is one of the common psychiatric disorders, with a worldwide prevalence of around 16·2%, with multifactorial causality, but partially unknown pathophysiology. Depression likely involves, at a molecular and cellular level, dysfunctions of critical neurotrophic, cellular plasticity and resilience pathways and neuroprotective processes.

In context to Neurotropic hypothesis, in depression there is reduction in Neurotrophins (NTs), which impairs the pruning of the neural network, alters neural plasticity, and impacts negatively on the structural and functional processes within the limbic system. NTs in general and Brain Derived Neurotrophic Factor (BDNF) in particular modulate depressive behavior and the response to antidepressant treatment, in part through the regulation of synaptic plasticity, synaptogenesis, and neurogenesis. Major neurotrophins like nerve growth factor (NGF), brain-derived neurotrophic factor (BDNF), neurotrophin-3 (NT-3) and neurotrophin-4/5 (NT-4/5) have been identified in context to nervous system functioning.

Previous studies have consistently proved the reduction in BDNF levels in patients with depression and antidepressants were found to increase BDNF protein levels with re-establishment of normative cortical networks in different areas of hippocampus. Recent studies have provided important links between the neurobiological characteristics of depression and NGF. Animal studies have revealed decreasing levels of NGF in specific brain areas of different mouse models, including anxiety vulnerability, stress-induced illness, and learned helplessness. In relation to the patients with depression, NGF has been recognized as an important factor in modulating their altered or dysfunctional hypothalamic-pituitary-adrenal (HPA) axis. Previous studies have compared the differences in peripheral NGF levels in patients with depression and healthy controls, others have investigated the effect of different treatments on their levels. The results have been conflicting in relation to NGF levels results before and after antidepressant treatment in patients with depression, thus, necessitating the need for further research in this area.

Studies related to NT-3 levels in unipolar depression is limited, when researchers have reported of increased CSF levels of NT-3 in elderly depressed patients and increased serum NT-3 levels in the depressive phase of Bipolar disorder. Lower level of neurotrophins like BDNF, but higher level of NT-3, have been found in depressed patients with schizophrenia. NT-4 has been a potential candidate neurotropic factor for research in patients with mood disorder. Studies have reported of increased serum NT-4 levels in the depressive phase of Bipolar disorder, when others have found the increase in serum NT-4 levels in both the depressive and manic phases of the illness. Contrastingly, studies have also found reduction in NT-4 levels in the manic phase of Bipolar disorder.

The literature search clearly reveals the lack of studies or inconsistent findings in relation to the role of major NTs like NGF, Neurotrophin-3, and Neurotrophin-4 in unipolar depression. It will be worth studying the changes in these NTs in depression and the effect of various antidepressants on their levels, this can help us in understanding the caveats in pathophysiology of depression better, which can have future treatment implications.

The aim of the present study will be to observe the changes in the NTs like Nerve growth factor, Neurotrophin-3, and Neurotrophin-4 in patients with depression and study the effect of various antidepressants like Sertraline (SSRI), Dosulepin (TCA), and Venlafaxine (SNRI) on their levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of Depressive episode (Single episode or recurrent) (by ICD-10 DCR) without psychotic symptoms.
* Patients aged 18-65 years, of either sex.
* Patients with baseline score > 7 on the Montgomery-Asberg Depression Rating Scale (MADRS).
* Treatment naïve or patients who had not taken any treatment for at least 4 weeks before inclusion.

Exclusion Criteria:

* Patients with Depressive episode (by ICD-10 DCR) with psychotic symptoms.
* Patients with Bipolar depression or with Persistent mood disorder (Dysthymia/ Cyclothymia)
* Patients who are already under treatment for the presenting conditions.
* Previous history of refractoriness to SSRI, TCA, or SNRI.
* Patients with comorbid substance abuse or history of organicity
* Patients with history of major medical or neurological illness.
* Pregnant and nursing women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with depression with or without somatic syndrome attending the outpatient department of Psychiatry, AIIMS, Bhubaneswar.
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change in serum nerve growth factor from baseline over 6 weeks | Baseline and 6 weeks
  ELISA

SECONDARY OUTCOMES:
Change in serum neurotrophin 3 from baseline over 6 weeks | Baseline and 6 weeks
  ELISA
Change in serum neurotrophin 4 from baseline over 6 weeks | Baseline and 6 weeks
  ELISA
Change in severity of symptoms of depression from baseline over 6 weeks | Baseline and 6 weeks
  Montgomery-Åsberg Depression Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: BISWA R MISHRA, MD, Principal Investigator — AIIMS, BHUBANESWAR
Locations (1):
- Dept of Psychiatry, Aiims, Bhubaneswar, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lee BH, Kim H, Park SH, Kim YK. Decreased plasma BDNF level in depressive patients. J Affect Disord. 2007 Aug;101(1-3):239-44. doi: 10.1016/j.jad.2006.11.005. Epub 2006 Dec 13. PMID 17173978
- [Result] Jiang C, Salton SR. The Role of Neurotrophins in Major Depressive Disorder. Transl Neurosci. 2013 Mar 1;4(1):46-58. doi: 10.2478/s13380-013-0103-8. PMID 23691270
- [Result] Chen B, Dowlatshahi D, MacQueen GM, Wang JF, Young LT. Increased hippocampal BDNF immunoreactivity in subjects treated with antidepressant medication. Biol Psychiatry. 2001 Aug 15;50(4):260-5. doi: 10.1016/s0006-3223(01)01083-6. PMID 11522260
- [Result] Chen YW, Lin PY, Tu KY, Cheng YS, Wu CK, Tseng PT. Significantly lower nerve growth factor levels in patients with major depressive disorder than in healthy subjects: a meta-analysis and systematic review. Neuropsychiatr Dis Treat. 2015 Apr 1;11:925-33. doi: 10.2147/NDT.S81432. eCollection 2015. PMID 25897228
- [Result] Liu X, Zhang T, He S, Hong B, Peng D, Su H, Li F, Tang Y, Lin Z, Fang Y, Jiang K. Nerve growth factor variations in patients with mood disorders: no changes in eight weeks of clinical treatment. Neuropsychiatr Dis Treat. 2014 May 15;10:835-40. doi: 10.2147/NDT.S62741. eCollection 2014. PMID 24868159
- [Result] Hock C, Heese K, Muller-Spahn F, Huber P, Riesen W, Nitsch RM, Otten U. Increased cerebrospinal fluid levels of neurotrophin 3 (NT-3) in elderly patients with major depression. Mol Psychiatry. 2000 Sep;5(5):510-3. doi: 10.1038/sj.mp.4000743. PMID 11032384
- [Result] Loch AA, Zanetti MV, de Sousa RT, Chaim TM, Serpa MH, Gattaz WF, Teixeira AL, Machado-Vieira R. Elevated neurotrophin-3 and neurotrophin 4/5 levels in unmedicated bipolar depression and the effects of lithium. Prog Neuropsychopharmacol Biol Psychiatry. 2015 Jan 2;56:243-6. doi: 10.1016/j.pnpbp.2014.09.014. Epub 2014 Oct 5. PMID 25290636
- [Result] Walz JC, Magalhaes PV, Giglio LM, Cunha AB, Stertz L, Fries GR, Andreazza AC, Kapczinski F. Increased serum neurotrophin-4/5 levels in bipolar disorder. J Psychiatr Res. 2009 Apr;43(7):721-3. doi: 10.1016/j.jpsychires.2008.10.005. Epub 2008 Dec 10. PMID 19081579
- [Result] Barbosa IG, Morato IB, Huguet RB, Rocha FL, Machado-Vieira R, Teixeira AL. Decreased plasma neurotrophin-4/5 levels in bipolar disorder patients in mania. Braz J Psychiatry. 2014 Oct-Dec;36(4):340-3. doi: 10.1590/1516-4446-2014-1380. Epub 2014 Jul 29. PMID 25076171
- [Result] Williams JB, Kobak KA. Development and reliability of a structured interview guide for the Montgomery Asberg Depression Rating Scale (SIGMA). Br J Psychiatry. 2008 Jan;192(1):52-8. doi: 10.1192/bjp.bp.106.032532. PMID 18174510